CLINICAL TRIAL: NCT07268820
Title: A Multicenter, Double-blind, Randomized, Investigator-initiated Trial to Evaluate the Degree of Symptom Relief of Zastaprazan and Esomeprazole in Patients With Erosive Reflux Disease With Night-time Heartburn Symptoms
Brief Title: Heartburn, Gastroesophageal Reflux Disease
Acronym: GERD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Byung-Wook Kim, Professor, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: JL-JAQ-402
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zastaprazan (Experimental): Zastaprazan 20 mg, once daily, preferably administered orally in the morning before breakfast for four weeks
  Interventions: Drug: Zastaprazan
- Esomeprazole (Active Comparator): Esomeprazole 40 mg, once daily, preferably administered orally in the morning before breakfast for four weeks
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Zastaprazan — Participants in this arm will receive zastaprazan. This group serves as the experimental treatment group exploratorily evaluating drug for GERD.
  Other Names: P-CAB
  Arms: Zastaprazan
Drug: Esomeprazole — Participants in this arm will receive esomeprazole. This group serves as the active comparator treatment group exploratorily evaluating drug for GERD.
  Other Names: PPI
  Arms: Esomeprazole

SUMMARY:
Gastroesophageal reflux disease (GERD) is a condition caused by the reflux of stomach contents into the esophagus, presenting with typical symptoms such as heartburn and acid regurgitation.

GERD is a chronic condition that affects quality of life, and patients with this condition are known to have a lower quality of life compared to healthy individuals. In particular, nocturnal heartburn can lead to sleep deprivation and affect daily life, as well as overall quality of life.

This study aims to evaluate the efficacy of alleviating nocturnal heartburn symptoms in patients with erosive reflux disease (ERD).

DETAILED DESCRIPTION:
This multicenter, double-blind, randomized, active-controlled Phase 4 study aims to exploratorily evaluate the comparative effects and safety of zastaprazan 20 mg and esomeprazole 40 mg in subjects with gastroesophageal reflux disease.

ELIGIBILITY:
Inclusion Criteria:

1. Korean adults aged 19 years or older as of the date of written consent
2. Those diagnosed with erosive gastroesophageal reflux disease based on upper gastrointestinal endoscopy (EGD)
3. Those who reported nighttime heartburn for more than 3 months at the time of screening (Visit 1)
4. Those who voluntarily decided to participate and provide written informed consent

Exclusion Criteria:

1. Those who cannot undergo upper gastrointestinal endoscopy (EGD)
2. Individuals with a history of drug or alcohol abuse (within the past year)
3. Individuals who have received other investigational products within one month prior to the screening visit (Visit 1)
4. In addition to the above, individuals with clinically significant findings that the investigator deems medically inappropriate for the present study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants without sleep disturbance related to nighttime heartburn during the last 7 days | Week 2
  This measure is based on participant-reported information collected by subject diary during the study and reflects whether sleep disturbance related to heartburn was noted over the period evaluated. Symptom severity ranges from 0 to 4, with higher scores indicating worse sleep disturbance.

SECONDARY OUTCOMES:
Proportion of participants without sleep disturbance related to nighttime heartburn during the last 7 days | Week 4
  This measure is based on participant-reported information collected by subject diary during the study and reflects whether sleep disturbance related to heartburn was noted over the period evaluated. Symptom severity ranges from 0 to 4, with higher scores indicating worse sleep disturbance.
Mean change from baseline in Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) score | Baseline, Week 2, Week 4
  The change from baseline in GERD-HRQL scores, evaluated at Weeks 2 and 4 during the treatment period. The GERD-HRQL uses item scores ranging from 0 to 5, with higher scores indicating more severe symptoms.
Mean change from baseline in Gastrointestinal Symptom Rating Scale (GSRS) score | Baseline, Week 2, Week 4
  The GSRS assesses gastrointestinal symptoms across multiple domains, with each item scored on a 1 to 7 scale, where higher scores indicate more severe symptoms.
Change from baseline in Gastroesophageal Reflux Disease Questionnaire (GerdQ) score | Baseline, Week 2, Week 4
  The GerdQ evaluates symptoms using ordinal item scores; for heartburn and acid regurgitation items, higher scores indicate more frequent symptoms; each item is scored on a 0 to 3 scale based on symptom frequency over the previous week, with reverse scoring applied to upper stomach pain and nausea items.

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Korea University Ansan Hospital, Ansan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Chilgok
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon
  - Chonnam National University Hospital, Gwangju
  - Catholic University of Korea, Incheon ST. Mary's Hospital, Incheon
  - Gangnam Severance Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No